CLINICAL TRIAL: NCT05249010
Title: The Effect of Moxibustion on the Meridian: A Prospective, Crossover Designed, Observational Study
Brief Title: The Effect of Moxibustion on the Meridian
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101924A3
Record Dates: First submitted 2022-01-28; First posted 2022-02-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-01

CONDITIONS: Acupuncture; Moxibustion
MeSH Terms: interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acupuncture and moxibustion group: The investigators intend to recruit 30 participants who receive acupuncture and then measure the VAS and electric characteristic by the semiconductor analyzer Agilent B1500A first. The investigators add the burned moxa on the acupuncture as a method for moxibustion, and then measure the VAS and electric characteristic again.
  Interventions: Procedure: acupuncture and moxibustion

INTERVENTIONS:
Procedure: acupuncture and moxibustion — Participants receive acupuncture and then measure the VAS and electric characteristic by the semiconductor analyzer Agilent B1500A first. The investigators add the burned moxa on the acupuncture as a method for moxibustion, and then measure the VAS and electric characteristic again.

SUMMARY:
The purpose of this study is to combine the Chinese medicine and physics, using acupuncture to conduct electrical measurement, and to understand the effects of moxibustion on meridian.

DETAILED DESCRIPTION:
Moxibustion is a traditional Chinese medicine, which use the burned moxa to generate warmth on the human's local skin and then exerts a therapeutic effect. Research found that moxibustion has effect on analgesic and anti-inflammation, which can be applied on myofascial pain, insomnia, osteoarthritis, osteoporosis, cancer related fatigue, irritable bowel disease etc.. Although research reveal that moxibustion can treat these diseases probably by effect on analgesic and anti-inflammation, the mechanism of moxibustion is still not clear.

In modern study, the meridian has electric characteristic and the therapeutic effect of acupuncture may be related to the electricity resulting by acupuncture manipulation. However, there is no study to investigate the electric effect of moxibustion on the meridian. In our study, the investigators applied the semiconductor analyzer Agilent B1500A to investigate the electric characteristic of meridians and visual analogue scale (VAS) before and after moxibustion, which may provide another vision on moxibustion in the future.

The investigators intend to recruit 30 healthy participants with age more than 20 years old to participate this study. The participants receive acupuncture and then measure the VAS and electric characteristic by the semiconductor analyzer Agilent B1500A immediately(baseline data). The investigators add the burned moxa on the acupuncture as a method for moxibustion. After the moxa burned out, the investigators measure the VAS and electric characteristic immediately again(post moxibustion data). The investigators will use paired t test and repeated measure two ways ANOVA to compare the VAS and electricity of baseline data and post moxibustion data in each participant.

The purpose of this study is to combine the Chinese medicine and physics, using acupuncture to conduct electrical measurement, and to understand the effects of moxibustion on meridian.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years old
* agree to the informed consent

Exclusion Criteria:

* under 20 years old
* pregnant or breast-feeding women
* those with an empty stomach before the study
* a tendency toward bleeding with thrombocytopenia or history of platelets < 20000 or a user of an anti-platelet drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from those considered healthy and at least 20 years old who agreed to the informed consent. The exclusion criteria for this study were: those under 20 years old, pregnant or breast-feeding women, those with an empty stomach before the study, a tendency toward bleeding with thrombocytopenia or platelets < 20000 or a user of an anti-platelet drug.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change of visual analogue scale (VAS), score from 0 to 10, the lower score means less pain while the higher score means more pain. | through study completion, an average of 90 minutes
  The investigators measure visual analogue score immediately after intervention of acupuncture (baseline data) and moxibustion (post moxibustion data) respectively.
  Measured time baseline data: immediately after acupuncture post moxibustion data: immediately after moxa burned out (10 minutes)
The change of electric current | through study completion, an average of 90 minutes
  Agilent B1500A is a device that can measure the electric current after acupuncture and moxibustion. The investigators measure the electric current after intervention of acupuncture (baseline data) and moxibustion (post moxibustion data) respectively.
  Measured time:
  baseline data: immediately after acupuncture post moxibustion data: immediately after moxa burned out (10 minutes)
The change of voltage | through study completion, an average of 90 minutes
  Agilent B1500A is a device that can measure the voltage after acupuncture and moxibustion. The investigators measure the voltage after intervention of acupuncture (baseline data) and moxibustion (post moxibustion data) respectively.
  Measured time:
  baseline data: immediately after acupuncture post moxibustion data: immediately after moxa burned out (10 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chiang Hung, Professor, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Sun Yat-Sen University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He XR, Wang Q, Li PP. Acupuncture and moxibustion for cancer-related fatigue: a systematic review and meta-analysis. Asian Pac J Cancer Prev. 2013;14(5):3067-74. doi: 10.7314/apjcp.2013.14.5.3067. PMID 23803081
- [Background] Lim MY, Huang J, Zhao B. Standardisation of moxibustion: challenges and future development. Acupunct Med. 2015 Apr;33(2):142-7. doi: 10.1136/acupmed-2014-010688. Epub 2014 Dec 15. PMID 25510253
- [Background] Hung YC, Chen WC, Chang TC, Zheng HX, Liu YW, Tan YF, Lin SK, Lu YH, Hu WL, Tsai TM. Meridian study on the response current affected by electrical pulse and acupuncture. Nanoscale Res Lett. 2020 Jul 10;15(1):146. doi: 10.1186/s11671-020-03373-2. PMID 32651748